CLINICAL TRIAL: NCT05290012
Title: The Effect of Dark Chocolate Consumption on Blood Parameters in Healthy Adult Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ETK00-2020-0283
Record Dates: First submitted 2022-01-21; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-01

CONDITIONS: Cardiovascular Diseases
Keywords: Chocolate; Cacao; Cholesterol; Blood Glucose; Blood Pressure
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dark Chocolate (Experimental): Participants consumed 18 grams of dark chocolate (36 g/day, 400 mg/day of flavanols) twice daily.
  Interventions: Other: Dark Chocolate
- Control (No Intervention): No intervention was made

INTERVENTIONS:
Other: Dark Chocolate — A daily consumption of 36 g dark chocolate (400 mg/day flavanol) was made. No Cocoa/chocolate product was consumed other than the intervention product.
  Arms: Dark Chocolate

SUMMARY:
In healthy individuals, the effect of regular dark chocolate consumption for 4 weeks on blood lipid parameters such as; total cholesterol, LDL cholesterol, HDL cholesterol and triglyceride levels, in addition to fasting blood glucose, HbA1c, CRP levels and blood pressure was investigated.

DETAILED DESCRIPTION:
Recent studies have shown that dark chocolate consumption may have a positive effect on cardiovascular risk markers.The aim of this study is to investigate the effect of regular consumption of dark chocolate (36 g/day) on biochemical blood parameters in healthy individuals. A total of 37 healthy individuals completed the study conducted in this direction. Participants were randomly divided into two groups as dark chocolate group (n=17) and control group (n=20). While the dark chocolate group consumed 36 g/day (400 mg/day flavanol) dark chocolate for 4 weeks, the control group did not receive any intervention. At the end of the study, the anthropometric measurements of the individuals were evaluated. Blood lipid profile, fasting blood glucose, HbA1c, CRP levels, systolic blood pressure and diastolic blood pressure measurements were investigated.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m2
* Systolic blood pressure <140 mmHg and/or diastolic blood pressure <90 mmHg

Exclusion Criteria:

* Individuals with any diagnosed chronic or acute illness
* Individuals diagnosed or in contact with Covid-19
* Individuals with allergies to cocoa/chocolate products
* Individuals in the process of losing weight
* Individuals with smoking and alcohol consumption
* Individuals taking medication or vitamin/mineral supplements
* Individuals doing heavy physical activity
* Individuals who regularly consume cocoa/chocolate products for the last 1 month (> 3 days a week)
* Pregnant or lactating women were excluded from the study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Change in serum lipid levels from baseline with dark chocolate consumption at 4 weeks. | Baseline and Week 4
  Serum lipid levels (total cholesterol, LDL cholesterol, HDL cholesterol and triglyceride) were measured by taking blood samples from individuals at the beginning and end of the study. Differences in blood lipid variables were analyzed using the Statistical Package for Social Sciences (SPSS) 24.0 program. Change = (Baseline serum lipid levels-Week 4 serum lipid levels)
Change in glycemic parameters from baseline with dark chocolate consumption at 4 weeks. | Baseline and Week 4
  At the beginning and end of the study, blood samples were taken from the individuals and their HbA1c and fasting blood glucose levels were measured. Differences in glycemic variables were analyzed using the Statistical Package for Social Sciences (SPSS) 24.0 program. Change = (Baseline glycemic parameters-Week 4 glycemic parameters)
Change in CRP levels from baseline with dark chocolate consumption at 4 weeks. | Baseline and Week 4
  At the beginning and end of the study, blood samples were taken from the individuals and their CRP (C-reactive protein) levels were measured. Differences in the CRP variable were analyzed using the Statistical Package for Social Sciences (SPSS) 24.0 program. Change = (Baseline CRP levels-Week 4 CRP levels)
Change in blood pressure from baseline with dark chocolate consumption at week 4. | Baseline and Week 4
  At the beginning and end of the study, the blood pressure (systolic blood pressure and diastolic blood pressure) measurements of the individuals were measured with the Nimo LD-520 digital blood pressure device. Change = (Baseline blood pressure-Week 4 blood pressure)

SECONDARY OUTCOMES:
Change in body weight from baseline with dark chocolate consumption at week 4. | Baseline and Week 4
  The body weight (kg) of the subjects was measured at the beginning and end of the study. The measurement was made with Tanita-BC-601. Change = (Baseline body weight-Week 4 body weight)
Change in BMI from baseline with dark chocolate consumption at week 4. | Baseline and Week 4
  The body mass index (BMI) of individuals at the beginning and end of the study was measured using mathematical calculation (weight/height squared; in kilograms per square metre).Change = (Baseline BMI-Week 4 BMI)
Change in body fat percentage from baseline with dark chocolate consumption at week 4. | Baseline and Week 4
  Body fat percentage (%) of individuals was measured at the beginning and end of the study. The measurement was made with Tanita BC-601. Change = (Baseline body fat percentage-Week 4 body fat percentage)
Change in waist circumference from baseline with dark chocolate consumption at week 4. | Baseline and Week 4
  At the beginning and end of the study, the waist circumference (cm) of the individuals (midway between the rib cage and the iliac crest) was measured using a flexible tape measure. Change = (Baseline waist circumference-Week 4 waist circumference)

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Küçükyılmaz, Principal Investigator — Eastern Medittanean University
Locations (1):
- Kübra Küçükyılmaz, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided